CLINICAL TRIAL: NCT04625816
Title: Comparison of Core Muscle Asymmetry Using Spine Balance 3D in Patients With Arthroscopic Shoulder Surgery: A STROBE-compliant Cross-sectional Study
Brief Title: Comparison of Core Muscle Asymmetry Using Spine Balance 3D in Patients With Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Principal Investigator, Sahmyook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020117HR
Record Dates: First submitted 2020-11-01; First posted 2020-11-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Muscle Disorder; Postoperative Pain; Shoulder Injuries; Immobilization; Asymmetric Limb Muscle Stiffness
MeSH Terms: conditions — Muscular Diseases; Pain, Postoperative; Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroscopic shoulder surgery patients (Experimental)
  Interventions: Device: whole body tilt device (Spine Balance 3D)

INTERVENTIONS:
Device: whole body tilt device (Spine Balance 3D) — The symmetry of the deep muscle was evaluated using a whole body tilt device (Spine Balance 3D, Cyber Medic Co., Ltd., Korea). Spine Balance 3D can evaluate the maintenance strength and maximum strength of the core muscles, and perform a personalized core muscle training program based on the evaluated results.

SUMMARY:
This study is an observational cross-sectional study. Post-operative patients need an immobilization period for a certain period of time after surgery. Kinetic chain changes due to immobilization can affect the symmetry of the core muscle. Therefore, in this study, core muscle asymmetry (CMA) is measured using a whole body tilt device for inpatients who have undergone arthroscopic shoulder surgery. We would like to make a clinical suggestion for post-operative rehabilitation by identifying the characteristics of CMA according to the left or right site.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic shoulder surgery
* limit of motion due to shoulder pain

Exclusion Criteria:

* orthopedic surgery or other medical history in the lower extremities
* neurological history or are taking related medications
* chronic headache or disease related to the inner ear
* cardiovascular disease that may affect balance ability or take related medications
* acute dizziness
* when performing other balance training

Ages: 26 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
direction core muscle ratio (DCMR) | 1 Day
  DCMR was calculated as a percentage of time located in each direction.
core muscle state ratio (CMSR) | 1 Day
  CMSR was calculated as a percentage of the value compared to the reference data of healthy adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
I plan to decide after the study is over.